CLINICAL TRIAL: NCT05807490
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED, PARALLEL STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF MULTIPLE ASCENDING ORAL DOSES OF PF-07328948 IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Learn How Different Amounts of the Study Medicine Called PF-07328948 Are Tolerated and Act in the Body in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C4921002; 2023-509054-54-00 (Other: CTIS (EU))
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: PF-07328948

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- PF-07328948 and Placebo (Cohort 1) (Experimental): Dose level 1: Multiple dose administration of PF-07328948 and placebo over 14 days in healthy participants; 8 participants will receive PF-07328948 and 2 will receive placebo
  Interventions: Drug: PF-07328948; Drug: Placebo
- PF-07328948 and Placebo (Cohort 2) (Experimental): Dose level 2: Multiple dose administration of PF-07328948 and placebo over 14 days in healthy participants; 8 participants will receive PF-07328948 and 2 will receive placebo
  Interventions: Drug: PF-07328948; Drug: Placebo
- PF-07328948 and Placebo (Cohort 3) (Experimental): Dose level 3: Multiple dose administration of PF-07328948 and placebo over 14 days in healthy participants; 8 participants will receive PF-07328948 and 2 will receive placebo
  Interventions: Drug: PF-07328948; Drug: Placebo
- PF-07328948 and Placebo (Cohort 4) (Experimental): Dose level 4: Multiple dose administration of PF-07328948 and placebo over 14 days in healthy participants; 8 participants will receive PF-07328948 and 2 will receive placebo
  Interventions: Drug: PF-07328948; Drug: Placebo
- PF-07328948 and Placebo (Cohort 5) (Experimental): Dose level 5: Multiple dose administration of PF-07328948 and placebo over 14 days in healthy participants; 8 participants will receive PF-07328948 and 2 will receive placebo
  Interventions: Drug: PF-07328948; Drug: Placebo
- PF-07328948 and Placebo (Cohort 10) (Experimental): Optional cohort - Multiple dose administration of PF-07328948 and placebo over 14 days in healthy Japanese participants; 5 participants will receive PF-07328948 and 1 will receive placebo
  Interventions: Drug: PF-07328948; Drug: Placebo
- PF-07328948 and Placebo (Cohort 7) (Experimental): Dose level 7: Multiple dose administration of PF-07328948 and placebo over 14 days in healthy participants; 8 participants will receive PF-07328948 and 2 will receive placebo
  Interventions: Drug: PF-07328948; Drug: Placebo
- PF-07328948 and Placebo (Cohort 8) (Experimental): Optional cohort - Dose level TBD. Multiple dose administration of PF-07328948 and placebo over 14 days in healthy participants; 8 participants will receive PF-07328948 and 2 will receive placebo
  Interventions: Drug: PF-07328948; Drug: Placebo
- PF-07328948 oral tablet and oral suspension (Cohort 11) (Experimental): Assessment of relative bioavailability PF-07328948 oral tablet compared to PF-07328948 oral suspension under fed and fasted condition; 12 participants will be enrolled, and 6 participants randomized to 1 of 2 sequences
  Interventions: Drug: PF-07328948
- PF-07328948 and Placebo (Cohort 6) (Experimental): Dose level 6: Multiple dose administration of PF-07328948 and placebo over 14 days in healthy participants; 8 participants will receive PF-07328948 and 2 will receive placebo
  Interventions: Drug: PF-07328948; Drug: Placebo
- PF-07328948 and Placebo (Cohort 9) (Experimental): Optional cohort - Dose level TBD. Multiple dose administration of PF-07328948 and placebo over 14 days in healthy participants; 8 participants will receive PF-07328948 and 2 will receive placebo
  Interventions: Drug: PF-07328948; Drug: Placebo

INTERVENTIONS:
Drug: PF-07328948 — PF-07328948 will be administered as oral suspensions every 12 hour (BID) over 14 days
  Arms: PF-07328948 and Placebo (Cohort 1)
Drug: Placebo — Placebo will be administered as oral suspensions BID over 14 days
  Arms: PF-07328948 and Placebo (Cohort 1)
Drug: PF-07328948 — PF-07328948 will be administered as oral suspensions daily (QD) over 14 days
  Arms: PF-07328948 and Placebo (Cohort 2)
Drug: Placebo — Placebo will be administered as oral suspensions QD over 14 days
  Arms: PF-07328948 and Placebo (Cohort 2)
Drug: PF-07328948 — PF-07328948 will be administered as oral suspensions every QD over 14 days
  Arms: PF-07328948 and Placebo (Cohort 3)
Drug: Placebo — Placebo will be administered as oral suspensions QD over 14 days
  Arms: PF-07328948 and Placebo (Cohort 3)
Drug: PF-07328948 — PF-07328948 will be administered as oral suspensions QD over 14 days
  Arms: PF-07328948 and Placebo (Cohort 4)
Drug: Placebo — Placebo will be administered as oral suspensions QD over 14 days
  Arms: PF-07328948 and Placebo (Cohort 4)
Drug: PF-07328948 — PF-07328948 will be administered as oral suspensions QD over 14 days
  Arms: PF-07328948 and Placebo (Cohort 5)
Drug: Placebo — Placebo will be administered as oral suspensions QD over 14 days
  Arms: PF-07328948 and Placebo (Cohort 5)
Drug: PF-07328948 — PF-07328948 will be administered as oral suspensions every 12 hour (BID) or everyday (QD) over 14 days
  Arms: PF-07328948 and Placebo (Cohort 10)
Drug: Placebo — Placebo will be administered as oral suspensions every 12 hour (BID) or everyday (QD) over 14 days
  Arms: PF-07328948 and Placebo (Cohort 10)
Drug: PF-07328948 — PF-07328948 will be administered as oral suspensions QD over 14 days
  Arms: PF-07328948 and Placebo (Cohort 7)
Drug: Placebo — Placebo will be administered as oral suspensions QD over 14 days
  Arms: PF-07328948 and Placebo (Cohort 7)
Drug: PF-07328948 — PF-07328948 will be administered as oral suspensions every 12 hour (BID) or daily (QD) over 14 days
  Arms: PF-07328948 and Placebo (Cohort 8)
Drug: Placebo — Placebo will be administered as oral suspensions every 12 hour (BID) or daily (QD) over 14 days
  Arms: PF-07328948 and Placebo (Cohort 8)
Drug: PF-07328948 — Single doses of PF-07328948 will be administered as oral suspension (single dose) and oral tablet (single dose) under fed and fasted condition
  Arms: PF-07328948 oral tablet and oral suspension (Cohort 11)
Drug: PF-07328948 — PF-07328948 will be administered as oral suspensions QD over 14 days
  Arms: PF-07328948 and Placebo (Cohort 6)
Drug: Placebo — Placebo will be administered as oral suspensions QD over 14 days
  Arms: PF-07328948 and Placebo (Cohort 6)
Drug: PF-07328948 — PF-07328948 will be administered as oral suspensions every 12 hour (BID) or daily (QD) over 14 days
  Arms: PF-07328948 and Placebo (Cohort 9)
Drug: Placebo — Placebo will be administered as oral suspensions every 12 hour (BID) or daily (QD) over 14 days
  Arms: PF-07328948 and Placebo (Cohort 9)
Drug: PF-07328948 — PF-07328948 will be administered as oral suspensions every 12 hour (BID) or daily (QD) over 14 days
  Arms: PF-07328948 and Placebo (Cohort 10)

SUMMARY:
This study has two parts: Part A and Part B.

The purpose of Part A of this study is to learn about the safety, tolerability, and how PF-07328948 is processed by the body when multiple doses of PF-07328948 are given to healthy participants.

The purpose of Part B of this study is to understand the amount of PF-07328948 that would be available in the body after taking a single pill. The amount will be compared to the amount of PF-07328948 in a suspension in healthy adults.

Part B will be conducted if the results of Part A support further study of PF-07328948.

The study is seeking participants who:

* are females who are not able to give birth to a child of 18 years of age or older.
* are males of 18 years of age or older.
* have a BMI of 20.0 to 35.0 kg/m2.
* have total body weight of more than 50 kg (110 lbs).

Participants in Part A will be randomly selected to receive either PF-07328948 or placebo (a pill that has no medicine in it).

Participants in Part B will receive PF-07328948 as suspension and tablet form, both taken by mouth after food or during fasting.

For a given participant in Part A, the total study is going to last up to about 12 weeks. This includes from the time of selection till the last follow-up phone call. The participants will be selected if they are fit for the study 28 days before the first dose of the study medicines. Participants who are selected will be admitted to the study site on Day -2 for around 19 days. Following discharge, participants will return for an on-site follow-up visit 7 to 10 days after receiving the final dose of the study medicine. The follow-up contact may be via a telephone call and will happen 28 to 35 days after the final dose of study medicine is given.

For a given participant in Part B, the total study is going to last up to about 10-12 weeks. Participants will stay overnight at the CRU for 23 days (Sequence 1) or 18 days (Sequence 2), starting with check-in. In Sequence 1, there will be a minimum of 10 days between doses in Period 1 and 2, and at least 7 days between doses in Period 2 and Period 3. In Sequence 2, there will be a minimum of 7 days between each dose.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants of non-childbearing potential and males must be 18 to 60 years of age for Part A and 18 to 65 years of age for Parts B at the time of signing the ICD, overtly healthy as determined by medical evaluation including medical history, physical exam, laboratory tests, and cardiac monitoring.
2. BMI of 20.0 to 35.0 kg/m2 and a total body weight >50 kg (110 lbs) for Part A. BMI of 17.5 to 35.0 kg/m2 and a total body weight >50 kg (110 lbs) for Part B.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
4. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological (including prothrombic/coagulopathic states), renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

   * Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
   * History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, HBcAb, or HCVAb. Hepatitis B vaccination is allowed.
2. Part B only: History of irregular bowel movements including irritable bowel syndrome or frequent episodes of diarrhea or constipation (defined as less than 1 bowel movement on average every 2 days) or lactose intolerance.
3. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to COVID-19 pandemic that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
4. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
5. Receipt of a COVID-19 vaccine within 7 days before screening or within 7 days before any visit in which a safety lab is planned. Vaccination with a COVID 19 vaccine that occurs greater than 7 days from either screening or any visit in which a safety lab is planned is permitted.
6. Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
7. Evidence of a prothrombotic state as evidenced by any of the following:

   * History of DVT, pulmonary embolism or arterial thrombosis.
   * Known genetic predisposition (Factor V Leiden, prothrombin G20210A, Protein C/S deficiency, antithrombin deficiency) based on medical history. Genetic testing at screening is not required.
   * ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test if deemed necessary:
   * presence of anti-phospholipid antibodies ("Positive" lab result for anticardiolipin, IgA, IgG or IgM)
   * Protein C activity < LLN of laboratory reference range
   * Protein S activity < LLN of laboratory reference range
   * Free Protein S antigen < LLN of laboratory reference range
   * Antithrombin activity < LLN of laboratory reference range
   * Positive test for APC resistance (Resistance Ratio < LLN of laboratory reference range)
   * Plasma fibrinogen > ULN of laboratory reference range
   * D-dimer ≥ 500 ng/ml (≥ 0.50 ug/ml)
8. A positive urine drug test.
9. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest.
10. Renal impairment as defined by an eGFR <75 mL/min/1.73m2 calculated using CKD EPI SCr formulas.
11. Standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF >450 ms, complete LBBB, signs of an acute or indeterminate age myocardial infarction, STT interval changes suggestive of myocardial ischemia, second- or third-degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the uncorrected QT interval is >450 ms, this interval should be rate corrected using the Fridericia method only and the resulting QTcF should be used for decision-making and reporting.
12. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

    * AST or ALT level ≥1.5× ULN;
    * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ULN.
13. Prior exposure to PF-07328948.
14. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit, or 3 ounces (90 mL) of wine).
15. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.
16. Use of tobacco or nicotine-containing products in excess of the equivalent of 5 cigarettes/day or 2 chews of tobacco/day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Part A: Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline up to 35 days after last dose of study intervention (approximately 11 weeks)
Part A: Number of Participants With Clinical Laboratory Abnormalities | Baseline up to 10 days after last dose of study intervention (approximately 7 weeks).
Part A: Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to 10 days after last dose of study intervention (approximately 7 weeks)
Part A: Number of Participants With Change From Baseline in Electrocardiogram (ECG) Findings | Baseline up to 10 days after last dose of study intervention (approximately 7 weeks)
Part A: Number of Participants With Change From Baseline in Physical Examination Findings | Baseline up to 10 days after last dose of study intervention (approximately 7 weeks)
Part A: Number of Participants With Cardiac Rhythms of Potential Clinical Concern Assessed By Telemetry | 0 to 8 hours post-dose on Day 1
Part A: Number of Participants With Cardiac Rhythms of Potential Clinical Concern Assessed By Telemetry | 0 to 8 hours post-dose on Day 14
Part B: Maximum Observed Plasma Concentration (Cmax) of PF-07328948 Tablet Formation and Oral Suspension | Predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours post dose on Day 1
Part B: Area Under the Plasma Concentration-time Curve from Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of PF-07328948 Tablet Formation and Oral Suspension | Predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours post dose on Day 1
Part B: Area Under the Plasma Concentration-time Curve from Time 0 to Extrapolated Infinite Time (AUCinf) of PF-07328948 Tablet Formation and Oral Suspension | Predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours post dose on Day 1

SECONDARY OUTCOMES:
Part A: Maximum Observed Plasma Concentration (Cmax) of PF-07328948 | predose, 0.25, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 38, and 72 hours post dose on Day 1
Part A: Maximum Observed Plasma Concentration (Cmax) of PF-07328948 | predose, 0.25, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 38, and 72 hours post dose on Day 14
Part A: Area Under the Plasma Concentration-Time Curve From Time 0 to Dosing Interval (tau) (AUCtau) of PF-07328948 | predose, 0.25, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 38, and 72 hours post dose on Day 1
Part A: Area Under the Plasma Concentration-Time Curve From Time 0 to Dosing Interval (tau) (AUCtau) of PF-07328948 | predose, 0.25, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 38, and 72 hours post dose on Day 14
Part A: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-07328948 | predose, 0.25, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 38, and 72 hours post dose on Day 1
Part A: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-07328948 | predose, 0.25, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 38, and 72 hours post dose on Day 14
Part A: Amount of PF-07328948 Excreted Unchanged in Urine Over the Dosing Interval Tau (Aetau) | On Day 14, urine collection for PK to occur over 0-tau, according to dosing frequency (ie, 0-12 hours for 12 hour dosing interval; 0-24 hours for 24 hour dosing interval)
Part A: Percentage of Dose of PF-07328948 Excreted Unchanged in the Urine Over the Dosing Interval Tau (Aetau%) | On Day 14, urine collection for PK to occur over 0-tau, according to dosing frequency (ie, 0-12 hours for 12 hour dosing interval; 0-24 hours for 24 hour dosing interval)
Part A: Renal Clearance of PF-07328948 | On Day 14, urine collection for PK to occur over 0-tau, according to dosing frequency (ie, 0-12 hours for 12 hour dosing interval; 0-24 hours for QD dosing interval)
Part B: Maximum Observed Plasma Concentration (Cmax) of PF-07328948 Tablet Formation Under Fasted and Fed Condition | predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours post dose on Day 1
Part B: Area Under the Plasma Concentration-time Curve from Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of PF-07328948 Tablet Formation Under Fasted and Fed Condition | predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours post dose on Day 1
Part B: Area Under the Plasma Concentration-time Curve from Time 0 to Extrapolated Infinite Time (AUCinf) of PF-07328948 Tablet Formation Under Fasted and Fed Condition | predose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours post dose on Day 1
Part B: Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline up to 35 days post dose of study intervention
Part B: Number of Participants With Clinical Laboratory Abnormalities | Baseline up to 4 days post dose of study intervention
Part B: Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to 4 days post dose of study intervention
Part B: Number of Participants With Change From Baseline in Electrocardiogram (ECG) Findings | Baseline up to 4 days post dose of study intervention
Part B: Number of Participants With Clinically-Significant Change From Baseline in Physical Examination Findings | Baseline up to 35 days post dose of study intervention
Part B: % of administered dose excreted in urine at each specified time interval | Days 1 to 11 at 24-hour intervals post-dose
Part B: Total % of PF-07328948 dose recovered in urine | Days 1 to 11 at 24-hour intervals post-dose
Part B: % of administered PF-07328948 dose excreted in feces at each specified time interval | Days 1 to 11 at 24-hour intervals post-dose
Part B: Total % of PF-07328948 dose recovered in feces | Days 1 to 11 at 24-hour intervals post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4921002